CLINICAL TRIAL: NCT07364370
Title: Myopia Progression Control Using Atropine 0.05% After Pediatric Cataract Surgery And Intraocular Lens Implantation Surgery: A Randomized Clinical Trial
Brief Title: Myopia Progression Control Using Atropine 0.05% After Pediatric Cataract Surgery And Intraocular Lens Implantation Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Awadein, Professor of Ophthalmology at Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-433-2025
Record Dates: First submitted 2026-01-05; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cataract; IOL Implantation; Myopia Progression
Keywords: pediatric cataract; iol; iol implantation; myopia
MeSH Terms: conditions — Intraocular Lymphoma; Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atropine (Experimental): Children receiving atropine 0.05% eye drops following IOL implantation. (as intervention)
  Interventions: Drug: Atropine Eye drops
- Control (No Intervention): Children receiving placebo eye drops following IOL implantation.

INTERVENTIONS:
Drug: Atropine Eye drops — Atropine eye drops, 0.05%, will be given following IOL implantation for a period of 12 months.
  Arms: Atropine

SUMMARY:
Myopic shift remains a debilitating and unpredictable adverse event following pediatric cataract surgery. While research exploring peripheral myopic defocus for post-cataract surgery myopia prevention shows promising results, the use of multifocal intra-ocular lenses (IOLs) cannot be used liberally in countries with high disease burden and challenged economies due to high price and decreased availability. To date there are no studies evaluating the use of topical atropine for the management of myopic shift following pediatric cataract surgery.

The investigators aim to explore the use of 0.05% topical atropine in the prevention and management of myopic shift following pediatric cataract surgery.

DETAILED DESCRIPTION:
Cataract is a leading cause of visual impairment in the pediatric age group, with an annual incidence of 1.8 to 3.6 per 10,000. The visual morbidity is not only due to media opacity caused by the cataracts, but also secondary to long lasting effects following cataract extraction, with timing and biometric aim of IOL implantation procedure presenting a unique challenge.

Normal ocular growth is characterized by axial length elongation along with corneal and lenticular flattening with a net refractive shift of approximately -0.9D. Cataract surgery in infants interrupts normal emmetropization of eyes and can lead to large myopic shift which may reach over 10 D.

Myopia is an epidemic with an estimated increase in prevalence to 50% by 2025. Rapidly progressing myopia significantly increases risk of permanent visual loss due to several ocular complications as maculopathy, retinal detachment and glaucoma.

Strategies for myopia control and prevention involve both optical and pharmacological measures, with atropine being a cornerstone in myopia management. Initially, it was believed that atropine limits myopia progression via blocking accommodation. Recently, however, it has been shown that atropine functions via a non-accommodative pathway. It is hypothesized that atropine exerts its action via regulation of dopamine release in retinal amacrine cells, which leads to reduction of rate of axial growth of eye. Another plausible mechanism is that up- and down-regulation of scleral muscarinic receptors influences scleral matrix deposition. Multiple low-dose concentrations have been studied, with older age and lower grades of myopia showing better response. Younger age requires the highest available concentration (0.05) to achieve adequate response.

While research exploring peripheral myopic defocus for post-cataract surgery myopia prevention shows promising results, the use of multifocal IOLs cannot be used liberally in countries with high disease burden and challenged economies due to high price and decreased availability. To date there are no studies evaluating the use of topical atropine for the management of myopic shift following pediatric cataract surgery.

The investigators aim to explore the use of 0.05% topical atropine in the prevention and management of myopic shift following pediatric cataract surgery.

ELIGIBILITY:
Inclusion criteria:

1. Children after IOL implantation (primary or secondary)
2. Age 1-7 years

Exclusion criteria:

1. Eyes with post-operative media opacity hindering adequate assessment of refraction
2. Eyes with complicated surgeries (e.g. vitreous loss, dropped lens matter requiring PPV, retinal detachment, etc)
3. Retinal pathologies
4. Glaucoma (congenital or secondary to surgery)
5. Anterior or posterior segment anomalies

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in spherical equivalent in diopters of each group. | Over a period of 12 months
  Spherical equivalent will be determined using auto-refractometer and/or manual retinoscopy. It will be reported in diopters (D).
Change in axial length in millimeters in each group. | 12 months
  Axial length will be measured using A-scan or optical biometry and will be reported in millimeters (mm).

SECONDARY OUTCOMES:
Rate of side-effects of atropine 0.05% eye drop use. | 12 months
  Rate of side-effects of atropine 0.05 eye drops will be reported as mydriasis leading to photophobia, blurring, and local allergic responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available upon request to rawan.m.hosny@students.kasralainy.edu.eg with strict patient anonymity ensured.
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT07364370/Prot_SAP_000.pdf